CLINICAL TRIAL: NCT05796518
Title: A Pilot Study to Examine Feasibility of a Patient Directed Tool to Assess Heart Health Among Endometrial Cancer Survivors
Brief Title: Feasibility of a Patient Directed Tool to Assess Heart Health Among Endometrial Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00095005; WFBCCC 99123 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Endometrial Cancer; Survivorship
Keywords: Heart health
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Endometrial cancer survivors presenting for post-treatment surveillance visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PREVENT - Cardiovascular Health Assessment Tool (Experimental): An adapted version of the PREVENT tool for endometrial cancer survivors will be used collect data during routine follow-up care for endometrial cancer that will yield a cardiovascular health score based on the Simple 7 risk factors (current smoking habits, body mass index, physical activity, diet, cholesterol, blood pressure and fasting plasma glucose).
  Interventions: Other: PREVENT Cardiovascular Health Assessment Tool; Other: Survey; Other: Interview Regarding Heart Health

INTERVENTIONS:
Other: PREVENT Cardiovascular Health Assessment Tool — Participants will access a heart health information visualization tool online using a personal device or a study tablet computer using their e-mail address to log-in. Investigators will review participant lab results specifically related to their cardiovascular health (e.g. blood pressure, cholesterol) in order to personalize the heart health tool for participants. A brief survey before and after use of the tool will also be completed by participants.
Other: Survey — A brief survey before and after use of the tool will also be completed by participants.
Other: Interview Regarding Heart Health — Participants will be asked questions related to their heart health.

SUMMARY:
Investigators are conducting this study to find out more about what heart health means to participants and how healthcare providers can best help to manage heart health. Participants will be asked to view an electronic tool designed to promote heart health awareness and help to manage heart health outside of the clinic. This study will provide important information to help investigators develop future programs that improve cancer patient's heart health after they complete their treatment.

DETAILED DESCRIPTION:
Primary Objective: The primary objective of this pilot study is to assess the feasibility of enrolling and completing the heart health assessment among endometrial cancer patients scheduled for routine follow-up care.

Secondary Objectives:

* To assess patient satisfaction with the tool.
* To identify the proportion of patients with non-ideal cardiovascular health scores who report initiating discussions regarding cardiovascular health during their routine oncology appointment.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a routine surveillance visit for pathologically confirmed stages I-IV endometrial cancer
* Greater than or equal to 3 months post-potentially curative cancer treatment
* Patients must be at least 18 years of age
* Have a working email address
* Comfortable reading medical information in English, as per self-report

Exclusion Criteria:

* Currently receiving treatment (e.g. radiation, chemotherapy, immunological treatments for endometrial cancer)
* Have a history of endometrial cancer recurrence
* Enrolled in hospice care or documentation of life expectancy < 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn E Weaver, PhD, MPH, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PREVENT - Cardiovascular Health Assessment Tool
Started | 44
Completed | 42
Not Completed | 2
Not completed — Were enrolled but did not complete the intervention | 2

BASELINE CHARACTERISTICS:
Arm/Group | PREVENT - Cardiovascular Health Assessment Tool
Number analyzed (Participants) | 42
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.5 [56.0 to 66.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 33
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants to Complete Intervention - Feasibility
Description: Feasibility will be defined from the number of participants who complete the web-based assessment using exact 95% binomial confidence intervals.
Time Frame: 6 months
Population: Out of the 44 participants enrolled only 42 complete the heart health assessment
Measure: Count of Participants; unit: Participants
Arm/Group | PREVENT - Cardiovascular Health Assessment Tool
Number analyzed (Participants) | 44
Participants | 42

2. Secondary Outcome: Number of Participants Stating Satisfaction With PREVENT Tool
Description: Patient satisfaction will be identified through post-visit survey with a 5-point Likert scale (strongly agree to strongly disagree) regarding liking the tool, helpfulness, ease of understanding and desire to use this tool with their oncologist. One-sample t-tests will be used to test whether the average response to each question is greater than 3.5 (with three denoting a neutral response). Wilcoxon signed rank tests will be used to compare cancer survivors' knowledge regarding their cardiovascular health risk factors and perceived importance of cancer and heart disease before and after using the cardiovascular risk visualization tool.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | PREVENT - Cardiovascular Health Assessment Tool
Number analyzed (Participants) | 42
Participants
  I am confident I understand my risk of heart disease: More Agreement | 4
  I am confident I understand my risk of heart disease: No Change | 36
  I am confident I understand my risk of heart disease: Less Agreement | 1
  I am confident I understand my risk of heart disease: Missing | 1
  I understand what steps I need to take to maintain or improve my heart health: More Agreement | 7
  I understand what steps I need to take to maintain or improve my heart health: No Change | 32
  I understand what steps I need to take to maintain or improve my heart health: Less Agreement | 1
  I understand what steps I need to take to maintain or improve my heart health: Missing | 2
  I plan to take steps to maintain or improve my heart health within the next year: More Agreement | 5
  I plan to take steps to maintain or improve my heart health within the next year: No Change | 34
  I plan to take steps to maintain or improve my heart health within the next year: Less Agreement | 1
  I plan to take steps to maintain or improve my heart health within the next year: Missing | 2
  Cancer poses a risk to my health: More Agreement | 6
  Cancer poses a risk to my health: No Change | 31
  Cancer poses a risk to my health: Less Agreement | 4
  Cancer poses a risk to my health: Missing | 1
  Heart disease poses a risk to my health: More Agreement | 8
  Heart disease poses a risk to my health: No Change | 22
  Heart disease poses a risk to my health: Less Agreement | 10
  Heart disease poses a risk to my health: Missing | 2
  I think it is important to talk to my oncology provider about heart health: More Agreement | 7
  I think it is important to talk to my oncology provider about heart health: No Change | 29
  I think it is important to talk to my oncology provider about heart health: Less Agreement | 4
  I think it is important to talk to my oncology provider about heart health: Missing | 2
  I think it is important to talk to my primary care provider about my heart health: More Agreement | 4
  I think it is important to talk to my primary care provider about my heart health: No Change | 26
  I think it is important to talk to my primary care provider about my heart health: Less Agreement | 9
  I think it is important to talk to my primary care provider about my heart health: Missing | 3
  Oncology providers should talk to their patients about their heart health: More Agreement | 7
  Oncology providers should talk to their patients about their heart health: No Change | 29
  Oncology providers should talk to their patients about their heart health: Less Agreement | 3
  Oncology providers should talk to their patients about their heart health: Missing | 3

3. Secondary Outcome: Number of Participants to Report Initiating Discussions Regarding Cardiovascular Health With Health Care Providers
Description: The initiation of discussions with participants' health care providers will largely be descriptive (using means as a measurement) to analyze this measure. Participants responded yes/no to the following discussions:
  1) Losing weight and maintaining a healthy body weight? 2) Quitting smoking, or staying smoke-free? 3) Controlling your blood pressure? 4) Controlling your cholesterol? 5) Controlling your glucose or hemoglobin A1c? 6) Any discussion regarding health with health care providers
Time Frame: 6 months
Population: Not all participants completed reported data on the health assessment tool
Measure: Count of Participants; unit: Participants
Arm/Group | PREVENT - Cardiovascular Health Assessment Tool
Number analyzed (Participants) | 42
Participants
  Losing weight and maintaining a healthy body weight?: number analyzed (Participants) | 35
  Losing weight and maintaining a healthy body weight?: Yes | 7
  Losing weight and maintaining a healthy body weight?: No | 28
  Quitting smoking, or staying smoke-free?: number analyzed (Participants) | 4
  Quitting smoking, or staying smoke-free?: Yes | 0
  Quitting smoking, or staying smoke-free?: No | 4
  Controlling your blood pressure?: number analyzed (Participants) | 39
  Controlling your blood pressure?: Yes | 11
  Controlling your blood pressure?: No | 28
  Controlling your cholesterol?: number analyzed (Participants) | 30
  Controlling your cholesterol?: Yes | 7
  Controlling your cholesterol?: No | 23
  Controlling your glucose or hemoglobin A1c?: number analyzed (Participants) | 31
  Controlling your glucose or hemoglobin A1c?: Yes | 9
  Controlling your glucose or hemoglobin A1c?: No | 22
  Any discussion regarding health with health care providers: Yes | 16
  Any discussion regarding health with health care providers: No | 26

ADVERSE EVENTS:
Time Frame: up to 3 months after using study tool
Arm/Group | PREVENT - Cardiovascular Health Assessment Tool
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT05796518/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT05796518/ICF_000.pdf